CLINICAL TRIAL: NCT00922376
Title: Assessment of the Clinical Efficacy and Acceptability of the Think Positive (T+) Diabetes Management System in Insulin Requiring Diabetes
Brief Title: Assessment of the Clinical Efficacy and Acceptability of Think Positive (T+) in Diabetes Management
Acronym: T+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College London Hospitals (Other)
Collaborators: University College, London (Other); Department of Health, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Justine Baron, Researcher, University College, London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/0201
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes (Insulin-requiring, Type 1 or Type 2)
Keywords: Diabetes; self- management; glycemic control; telehealth; mhealth
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- T+ Intervention (Active Comparator): The intervention group patients will use the T+ telemedicine application whilst completing repeated measures aiming to compare them to a control group receiving standard care.
  Interventions: Device: Mobile phone telehealth application: Think Positive (T+)
- Usual care (No Intervention): The control group will be receiving the standard care offered by the NHS to patients suffering from diabetes.

INTERVENTIONS:
Device: Mobile phone telehealth application: Think Positive (T+) — T+ consists of the Glucometer paired with a cradle that transmits via Bluetooth blood glucose results to a mobile phone. Data is stored and sent to a secure website. The website can be accessed by the patient as well as by health care providers (HCP). HCP can discuss data on the phone and make recommendations via text messages to patients. Visual feedback (graphs and statistics) illustrating recent blood sugar levels patterns is automatically and immediately sent to the patient when data is transferred from the T+ phone.
  Arms: T+ Intervention

SUMMARY:
New telemedicine systems have been designed to assist people suffering from diabetes in the management of their chronic disease. More recently the focus has been moving to portable systems equipped with Bluetooth. This study consists of evaluating an application called the Think Positive (T+) diabetes management software. It is a randomized controlled trial designed to compare, over a nine month period, a group of patients receiving usual care with a group of patients using the T+ system. The objectives of the study are to investigate the extent to which this telemedicine application helps patients control their blood sugar levels (HbA1c), as well as the extent to which its users consider it to be acceptable. The impact of its use on factors such as diabetes self-care, health status, quality of life, self-confidence in diabetes management, fear of hypoglycemia and illness representations will also be examined. Because of the supplementary real-time support and feedback that T+ offers, its use should lead to better outcomes in diabetes management than usual care does.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 and type 2 diabetes patients
* Insulin requiring patients
* Sufficiently fluent in english
* HbA1c > 7.5
* Last visit with Diabetes Specialist Nurse (DSN) < 12 months

Exclusion Criteria:

* Psychiatric disorders
* Poor vision or/and lack of manual dexterity
* Prior use of T+
* Participation in another ongoing trial
* Patients with antenatal/gestational
* Patients who are in transition between the children services and adult services Insulin pump users

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Blood sugar levels (HbA1c) | Baseline, 3 months, 9 months

SECONDARY OUTCOMES:
BMI | Baseline, 3 months, 9 months
Number of Hypoglycemic events | Baseline, 3 months, 9 months
Blood pressure | Baseline, 3 months, 9 months
Diabetes self-care | Baseline, 3 months, 9 months
Diabetes self- efficacy | Baseline, 3 months, 9 months
Quality of life | Baseline, 3 months, 9 months
Health status | Baseline, 3 months, 9 months
Illness representations | Baseline, 3 months, 9 months
User acceptability of T+ | 3 months, 9 months
Nurses' Perceptions of T+ | Baseline, 3 months, 9 months
Self efficacy in using T+ | 3 months, 9 months
Health care utilization | baseline, 3 months, 9 months
Self management | baseline, 3 months, 9 months
  2 subscales of the HeiQ questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London (UCL), London, United Kingdom

REFERENCES:
- [Background] Blake H. Mobile phone technology in chronic disease management. Nurs Stand. 2008 Nov 26-Dec 2;23(12):43-6. doi: 10.7748/ns2008.11.23.12.43.c6728. PMID 19093357
- [Background] Farmer A, Gibson OJ, Tarassenko L, Neil A. A systematic review of telemedicine interventions to support blood glucose self-monitoring in diabetes. Diabet Med. 2005 Oct;22(10):1372-8. doi: 10.1111/j.1464-5491.2005.01627.x. PMID 16176199
- [Background] Faridi Z, Liberti L, Shuval K, Northrup V, Ali A, Katz DL. Evaluating the impact of mobile telephone technology on type 2 diabetic patients' self-management: the NICHE pilot study. J Eval Clin Pract. 2008 Jun;14(3):465-9. doi: 10.1111/j.1365-2753.2007.00881.x. Epub 2008 Mar 24. PMID 18373577
- [Background] Jaana M, Pare G. Home telemonitoring of patients with diabetes: a systematic assessment of observed effects. J Eval Clin Pract. 2007 Apr;13(2):242-53. doi: 10.1111/j.1365-2753.2006.00686.x. PMID 17378871
- [Background] Kollmann A, Riedl M, Kastner P, Schreier G, Ludvik B. Feasibility of a mobile phone-based data service for functional insulin treatment of type 1 diabetes mellitus patients. J Med Internet Res. 2007 Dec 31;9(5):e36. doi: 10.2196/jmir.9.5.e36. PMID 18166525
- [Background] Wangberg SC, Arsand E, Andersson N. Diabetes education via mobile text messaging. J Telemed Telecare. 2006;12 Suppl 1:55-6. doi: 10.1258/135763306777978515. PMID 16884582
- [Derived] Baron J, Hirani S, Newman S. A mobile telehealth intervention for adults with insulin-requiring diabetes: early results of a mixed-methods randomized controlled trial. JMIR Res Protoc. 2015 Feb 26;4(1):e27. doi: 10.2196/resprot.4035. PMID 25803226